CLINICAL TRIAL: NCT03375957
Title: A Single-Site Study To Evaluate the Sensitization Potential of Topically Applied ATx201 in Healthy Human Volunteers
Brief Title: Sensitization Study of ATx201 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATx201-005
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Sensitivity, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ATx201 2% Gel (Experimental)
  Interventions: Drug: ATx201
- ATx201 4% Gel (Experimental)
  Interventions: Drug: ATx201
- ATx201 Gel Placebo (Placebo Comparator)
  Interventions: Drug: ATx201 Placebo Gel

INTERVENTIONS:
Drug: ATx201 — two hundred microliters (200 μL) of test article applied to the test site areas of the upper outer arms
  Arms: ATx201 2% Gel; ATx201 4% Gel
Drug: ATx201 Placebo Gel — two hundred microliters (200 μL) of placebo applied to the test site areas of the upper outer arms
  Arms: ATx201 Gel Placebo

SUMMARY:
This is a Phase I, single-site study to evaluate the sensitization potential of topically applied ATx201 GEL, 2% and 4%, along with a placebo control, in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Body Mass Index no less than 19.0 and no greater than 36.0 kg/m² (inclusive).
* Demonstrates a Fitzpatrick skin score of I - IV
* Female subjects must agree to use acceptable contraceptive methods from the Screening Visit through 90 days after the End of Study (EOS) Visit; or postmenopausal status with no menses for at least 1 year prior to the Screening Visit.
* Willing to refrain from excessive consumption of sodium in food or beverage 48 hours prior to Day 1 through EOS Visit.
* Willing to shower using the same non-medicated soap/cleansers, and abstain from excessive sun exposure (including tanning salons) from the Screening Visit through EOS Visit.

Exclusion Criteria:

* Reports a history of diabetes mellitus, clinically significant asthma (acceptable if no episode within 5 years prior to Day 1), or currently diagnosed with hypertension or circulatory disease.
* Reports use of any oral, nasal or topical corticosteroids, or oral or topical retinoids (other than Vitamin A at normal dietary amounts)
* Reports a significant history of allergy to soaps, lotions, emollients, ointments, creams, cosmetics, adhesives, or latex.
* Reports a history of significant skin conditions or disorders such as psoriasis, atopic dermatitis, etc.
* Reports a history of significant dermatologic cancers.
* Displays an obvious difference in skin color between upper arms or upper back or the presence of a skin anomaly
* Reports smoking or use of tobacco or nicotine delivery products within 14 days prior to Day 1 through EOS Visit.
* Presence of any clinically significant results from laboratory tests and vital signs assessments, as judged by the Investigator.
* A female who is pregnant, lactating, breastfeeding, or intends to become pregnant over the course of the study.
* Reports a history of drug or alcohol addiction or abuse within the past year.
* Reports having donated blood or plasma within 48 hours prior to Day 1 through EOS Visit.
* Subject exhibits excessive hair density on the upper arms or back such that patch adhesion could be compromised.
* Subject reports undergoing hair depilation (e.g. chemical, laser, physical) within 30 days prior to Day 1 through EOS Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Dermal Response Score | 21 days
  number of patients with a dermal response score of at least 2

SECONDARY OUTCOMES:
Dermal Response and Effects Score | 21 days
  number of patients with a dermal response and effects score of at least 3

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Director — CMO
Locations (1):
- Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No